CLINICAL TRIAL: NCT04601103
Title: 3M Oral Rinse Evaluation of Incidence and Patient Acceptance of Sloughing When Used With Sodium Lauryl Sulfate (SLS) Toothpastes
Brief Title: 3M Oral Rinse Incidence and Patient Acceptance of Sloughing When Used With Sodium Lauryl Sulfate (SLS) Toothpastes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device Deficiency
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EM-11-050043
Record Dates: First submitted 2020-10-13; First posted 2020-10-23 (Actual); Results first posted 2021-11-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Oral Mucosal Disorder

STUDY DESIGN:
Intervention Model Description: The study was designed as an imbalanced 2 Period Crossover Study. However, the study was terminated during the washout period and the results reported here reflect only the period 1 results.
Who Masked: Outcomes Assessor
Masking Description: Assessors did not know what toothpaste subjects used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Comparator: No SLS Toothpaste (Experimental): 3M Oral Rinse in combination with no SLS toothpaste (A)
  Interventions: Drug: No SLS toothpaste; Device: Anti-plaque
- Comparator: Medium SLS Toothpaste (Experimental): 3M Oral Rinse in combination with medium SLS toothpaste (B)
  Interventions: Drug: Medium SLS toothpaste; Device: Anti-plaque
- Comparator: High SLS Toothpaste (Experimental): 3M Oral Rinse in combination with high SLS toothpaste (C)
  Interventions: Drug: High SLS toothpaste; Device: Anti-plaque

INTERVENTIONS:
Drug: No SLS toothpaste — Toothpaste no Sodium Lauryl Sulfate
  Other Names: Sensodyne ProNamel Fresh Breath Toothpaste
  Arms: Comparator: No SLS Toothpaste
Drug: Medium SLS toothpaste — Less than or equal to X ppm Sodium Lauryl Sulfate
  Other Names: Clinpro Tooth Creme
  Arms: Comparator: Medium SLS Toothpaste
Drug: High SLS toothpaste — More than or equal to X ppm Sodium Lauryl Sulfate
  Other Names: Colgate Cavity Protection Toothpaste
  Arms: Comparator: High SLS Toothpaste
Device: Anti-plaque — Rinse prevents bacterial adherence to teeth
  Other Names: 3M Oral Rinse

SUMMARY:
The primary objective of this study is to evaluate the incidence of oral tissue sloughing through self-report by study subjects and by professional dental examinations.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the incidence of oral tissue sloughing through self-report by study subjects and by professional dental examinations. Adverse events will be tracked through study dental examinations and subject diaries with twice daily use of the 3M Oral Rinse used in combination with toothpaste containing one of three levels (no, medium, high) of Sodium Lauryl Sulfate (SLS).

Determine the subjects' acceptance of sloughing and/or other side effects

ELIGIBILITY:
Inclusion Criteria

1. Able to understand and willing to sign the informed consent;
2. Willing to agree to maintain confidentiality of the study and study materials;
3. 3M employee aged 18 years and older;
4. Willing to return to the study facility for scheduled study visits and recalls;
5. Agree not to use other oral hygiene products (non-study toothpaste, non-study toothbrush, mouth rinse, chewing gum);
6. Agree to the study instruction and schedule

   Exclusion Criteria:
7. A member of the Medical Clinical Affairs (MCA) staff or Panda product team for the device under investigation;
8. Have a dental appointment scheduled during study duration for professional cleaning;
9. Is pregnant, nursing, or planning to become pregnant within the study duration;
10. History of antibiotic therapy within the previous 30 days or have a condition that is likely to need antibiotic treatment over the course of the study (e.g., cardiac conditions requiring antibiotic prophylaxis such as heart murmurs, pacemakers, or prosthetic heart valves and prosthetic implants);
11. History of using a prescription antimicrobial mouth rinse during the past 3 months;
12. Currently taking medications which may alter gingival appearance/bleeding;
13. Currently using anticonvulsants, calcium channel blockers, or other medications with side effects known to impact oral health;
14. Participation in any other clinical study within the last 30 days;
15. Resides in the same household with a subject already enrolled in the study;
16. Known history of sensitivity to oral hygiene products;
17. Currently using tobacco products (cigarettes, chewing tobacco) or vaping products (ecigarettes);
18. History of diabetes;
19. Have removable partial/full dentures;
20. Have orthodontic appliances;
21. Have medical or oral conditions that may compromise the subject's safety or interfere with the conduct and outcome of the study;
22. Have known sloughing within the last 3 weeks;
23. Have dry mouth;
24. Have widespread caries or chronic neglect;
25. Have gross pathological changes of oral soft tissues;
26. Have advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive alveolar bone loss);
27. Unsuitable for enrollment in this study based on the professional opinion of the dental examiner based on the oral exam or other reasons not specified in the protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda C Coalwell, BA, Principal Investigator — 3M Health Care Business Group
Locations (1):
- 3M Health Care, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Comparator: No SLS Toothpaste: 3M Oral Rinse in combination with no SLS toothpaste (A)
  No SLS toothpaste: Toothpaste no Sodium Lauryl Phosphate
  Anti-plaque: Rinse prevents bacterial adherence to teeth
- Comparator: Medium SLS Toothpaste: 3M Oral Rinse in combination with medium SLS toothpaste (B)
  Medium SLS toothpaste: Less than or equal to X ppm Sodium Lauryl Phosphate
  Anti-plaque: Rinse prevents bacterial adherence to teeth
- Comparator: High SLS Toothpaste: 3M Oral Rinse in combination with high SLS toothpaste (C)
  High SLS toothpaste: More than or equal to X ppm Sodium Lauryl Phosphate
  Anti-plaque: Rinse prevents bacterial adherence to teeth
Period: Overall Study
Arm/Group | Comparator: No SLS Toothpaste | Comparator: Medium SLS Toothpaste | Comparator: High SLS Toothpaste
Started | 18 | 18 | 17
Completed | 0 | 0 | 0
Not Completed | 18 | 18 | 17
Not completed — Needed crown & cleaning | 0 | 0 | 1
Not completed — study was terminated | 18 | 18 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comparator: No SLS Toothpaste | Comparator: Medium SLS Toothpaste | Comparator: High SLS Toothpaste | Total
Number analyzed (Participants) | 18 | 18 | 17 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (10.3) | 39.7 (12.09) | 38.5 (11.82) | 40.5 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 9 | 31
  Male | 7 | 7 | 8 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 16 | 18 | 16 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 18 | 17 | 17 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 17 | 53
Number of Participants with Oral Tissue Sloughing at Baseline [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Oral Mucosal Exfoliation (Oral Sloughing)
Description: Percentage of participants who experienced oral sloughing as reported either by the subject or determined by the dental evaluator.
Time Frame: End of treatment (3 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Comparator: No SLS Toothpaste | Comparator: Medium SLS Toothpaste | Comparator: High SLS Toothpaste
Number analyzed (Participants) | 18 | 18 | 17
Participants | 15 | 14 | 13
Statistical Analysis 1: Comparison: Comparator: No SLS Toothpaste vs Comparator: Medium SLS Toothpaste vs Comparator: High SLS Toothpaste; Test type: Other — Generalized Fisher's Exact Test was used to detect an association between the 3 treatment groups and the incidence of sloughing; p = .916, Fisher Exact

2. Secondary Outcome: The Number of Participants With a Given Range of Average Oral Mucosal Sloughing Index Scores
Description: Average score based on the mean of sloughing scores over 12 intra-oral areas. The sloughing score uses a 6 point scale as follows: 0= no sloughing, 1=flecks of desquamation, 2=sheets of desquamation, 3=redness, not due to plaque, 4=erosion of mucosa, 5=ulcerated areas.
  The twelve intra-oral areas of the mouth are as follows: dorsal and ventral surfaces of the tongue, floor and roof of the mouth, right and left buccal mucosa, gingival tissue.
  (upper right, upper anterior, upper left, lower left, lower anterior, lower right)
Time Frame: Mid-Treatment (10 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Comparator: No SLS Toothpaste | Comparator: Medium SLS Toothpaste | Comparator: High SLS Toothpaste
Number analyzed (Participants) | 18 | 18 | 16
Participants
  0 no sloughing | 8 | 6 | 7
  (0.0, 0.5] | 9 | 8 | 6
  (0.5, 1.0] | 1 | 3 | 2
  (1.0, 1.5] | 0 | 0 | 1
  (1.5, 2.0] | 0 | 1 | 0

3. Secondary Outcome: The Number of Participants With a Given Range of Average Oral Mucosal Sloughing Index Scores.
Description: as for outcome 2
Time Frame: End of Treatment (3 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Comparator: No SLS Toothpaste | Comparator: Medium SLS Toothpaste | Comparator: High SLS Toothpaste
Number analyzed (Participants) | 18 | 18 | 16
Participants
  0 No sloughing | 6 | 9 | 7
  (0.0, 0.5] | 9 | 6 | 6
  (0.5, 1.0] | 3 | 2 | 2
  (1.0, 1.5] | 0 | 1 | 1

4. Other Pre Specified Outcome: The Number of Participants Reporting Their Acceptance Levels of Side Effects
Description: Subjects were questioned regarding how acceptable were your side effects. Using the following responses of: Completely unacceptable, somewhat unacceptable, somewhat acceptable, completely acceptable, did not experience side effects
Time Frame: End of Treatment (3 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Comparator: No SLS Toothpaste | Comparator: Medium SLS Toothpaste | Comparator: High SLS Toothpaste
Number analyzed (Participants) | 18 | 18 | 17
Participants
  Completely unacceptable | 2 | 1 | 2
  Somewhat unacceptable | 2 | 0 | 1
  Somewhat acceptable | 1 | 4 | 4
  Completely acceptable | 1 | 4 | 3
  Did not experience side effects | 12 | 9 | 7

ADVERSE EVENTS:
Time Frame: Within 3 weeks of starting treatment
Arm/Group | Comparator: No SLS Toothpaste | Comparator: Medium SLS Toothpaste | Comparator: High SLS Toothpaste
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 15/18 | 15/18 | 16/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comparator: No SLS Toothpaste (N=18) | Comparator: Medium SLS Toothpaste (N=18) | Comparator: High SLS Toothpaste (N=17)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Breath odor (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Buccal mucosal roughening (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Dysgeusia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3)
Mouth injury (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oral mucosal exfoliation (Gastrointestinal disorders) | 15 (15) | 14 (14) | 13 (13)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Tongue biting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue exfoliation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Device failure (Product Issues) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The major limitation with this study is that the sample size goal was not reached given the early termination during the washout period of a two-period crossover design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT04601103/Prot_SAP_000.pdf